CLINICAL TRIAL: NCT03511430
Title: Performance of a New Risk Score (SVEAT Index) to Identify Low-risk Patients Presenting to Emergency Department With Acute Chest Pain
Brief Title: "SVEAT" Chest Pain Scoring System
Status: Completed | Type: Observational
Sponsor: University of Nevada, Reno (Other)
Collaborators: Renown Regional Medical Center (Other)
Responsible Party: Principal Investigator, Chanwit Roongsritong, MD. FACC., University of Nevada, Reno
Other Study IDs: 986654
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Chest Pain
Keywords: Acute Coronary Syndrome; Heart Diseases; Cardiovascular Diseases; Vascular Diseases
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Heart Diseases; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational study to assess the efficacy of the newly developed SVEAT scoring system in identifying low-risk patients who may be eligible for early discharge. Various elements of clinical information including Symptoms, Vascular history, EKG, Age and Troponin values will be checked and entered on the scoring form to calculate the SVEAT risk score. Additionally, HEART score and TIMI risk score will be calculated for the same subjects.

The primary aim is to assess the positive and negative predictive values for the SVEAT index for cardiovascular events and compare it to the HEART and TIMI Scores.

DETAILED DESCRIPTION:
This is a prospective, observational study in patients presenting to the emergency department or admitted to clinical decision unit at Renown Regional Medical Center with a primary complaint of chest pain in a period of 12 months.

All patient >24 years will be recruited. Exclusion criteria include patients with clear-cut acute ST-segment elevation myocardial infarction, traumatic non-cardiac chest pain, life-expectancy less than 90 days, hemodynamic instability or inability to provide informed consent. Data and scores based on commonly known TIMI* risk score, HEART score and a newly developed SVEAT index ( Symptoms, Vascular disease, EKG, Age, Troponin) will be obtained by primary investigator trained physicians or advanced nurse practitioners as earliest as possible after their initial presentation. The care of the patients will be left to the discretion of the treating physician.

The outcome of each patient will be determined by either chart review, telephone contact or office visit as appropriate in 30 days post presentation. The sensitivity, specificity, positive and negative predictive value of SVEAT index will be calculated using standard statistical analysis. The receiver operating characteristic (ROC) curves of SVEAT index, TIMI risk score and HEART score will be generated and compared using commercially available software. P value of 0.05 or less will be considered statistically significant difference.

The primary hypothesis of the study is that scoring systems that better incorporate useful clinical information such as the SVEAT score may improve our ability to accurately identify low-risk acute chest pain patients presenting to the ED.

ELIGIBILITY:
Inclusion Criteria:

* Any patient > 24 years old presenting to the emergency room or admitted to the clinical decision unit with chest pain.

Exclusion Criteria:

* patient with clear-cut acute ST-segment elevation myocardial infarction, traumatic non-cardiac chest pain, life-expectancy less than 90 days, hemodynamic instability or inability to provide informed consent.

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient >24 years of age presenting to the emergency department or admitted to clinical decision unit at Renown Regional Medical Center with a primary complaint of chest pain.
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Occurence of MACE (Major Adverse Cardiac Events) | 30 days
  The number of subjects diagnosed with MACE (Acute Myocardial Infarction, Percutaneous Coronary Intervention, Coronary Artery Bypass Grafting, Significant stenosis with conservative therapy, Death)

CONTACTS AND LOCATIONS:
Overall Officials: Chanwit Roongsritong, MD, FACC, Principal Investigator — University of Nevada, Reno
Locations (1):
- Renown Regional Medical Center, Reno, Nevada, United States

REFERENCES:
- [Derived] Roongsritong C, Taha ME, Pisipati S, Aung S, Latt H, Thomas J, Namballa L, Al-Hasnawi HJ, Taylor MK, Gullapalli N. SVEAT Score, a Potential New and Improved Tool for Acute Chest Pain Risk Stratification. Am J Cardiol. 2020 Jul 15;127:36-40. doi: 10.1016/j.amjcard.2020.04.009. Epub 2020 Apr 20. PMID 32418720